CLINICAL TRIAL: NCT03516292
Title: Potential Biomarkers in the Study of Overactive Bladder in Women
Brief Title: Assessment of Potential Biomarkers in Women With Symptoms of Overactive Bladder and Pelvic Organ Prolapse
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Sofia Tsiapakidou, Principal Investigator, PhD Candidate, Resident Doctor in Obstetrics & Gynecology,, Aristotle University Of Thessaloniki
Other Study IDs: 411/29.03.2018
Record Dates: First submitted 2018-04-22; First posted 2018-05-04 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; biomarker; nerve growth factor; vaginal prolapse; urinary incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Hereditary Sensory and Autonomic Neuropathies; Uterine Prolapse; Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine sample of female patients with POP and POP with OAB
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OAB-POP group: As an Observational Case-Control Study, the participants will divided in two groups depending whether they suffer from overactive bladder symptoms or not. All participants will have POP.
  Interventions: Diagnostic Test: Urinary Nerve Growth Factor
- POP only group: As an Observational Case-Control Study, the participants will divided in two groups depending whether they suffer from overactive bladder symptoms or not. All participants will have POP.
  Interventions: Diagnostic Test: Urinary Nerve Growth Factor

INTERVENTIONS:
Diagnostic Test: Urinary Nerve Growth Factor — The subjective patient's discomfort regarding the vaginal prolapse problems and urinary incontinency symptoms will be assessed through the following questionnaires: (a) ICIQ-OAB (b) ICIQ FLUTS (c) ICIQ-VS. Determination of the bladder neck of urethra in midsagittal plane using a transvaginal two-dimensional ultrasound machine at lithotomy position in rest (point OA) and on Valsalva maneuver (point OB). Bladder Neck Mobility is defined as the difference from point OA to OB. BWT is determined and measured as the hypoechoic layer between two hyperechoic layers that is recognized as the urothelium and the perivesical tissue using a transvaginal two-dimensional ultrasound machine at lithotomy position. The measurement is performed with a bladder volume <30 ml and is taken place in 3 different bladder sites: (a) the thickest part of the bladder triangle, (b) the dome of the bladder in the midline, (c) the anterior wall of the bladder. NGF will be measured in urine sample.
  Other Names: Bladder Wall Thickness; Bladder Neck Mobility; Clinical Assessment of Subjective Vaginal and Urinary Symptoms

SUMMARY:
The objective of this study is to investigate the role of certain biomarkers in the initial assessment of women with overactive bladder (OAB). Nerve Growth Factor (NGF) levels, measured in urine samples, and bladder wall thickness (BWT), determined by two-dimensional transvaginal ultrasound, are two of those markers. The investigators hypothesize that the pre-operative determination of these biomarkers in women suffering from genital prolapse and overactive bladder could lead to a more accurate prognosis of the post-operative course of overactive bladder symptoms in women undergoing surgical treatment of prolapse.

DETAILED DESCRIPTION:
Pelvic organ prolapse Pelvic organ prolapse (POP) is a clinical condition that, although it is not life-threatening, significantly affects patients' quality of life. POP affects more than 30% of females in the general population. Among those, the majority is free of symptoms and do not need any medical assistance. However, according to US statistics, almost 20% of women will be candidates for some type of surgery to restore POP during their lifetime.

Urinary incontinence Urinary incontinence (UI) is used to describe any loss of urine through the urethra. It is a common patient complaint but not a specific disease. UI significantly affects patients' quality of life. UI is classified in 3 subtypes: stress UI (SUI) (loss of urine on effort, coughing etc.), urgency UI (UUI) (loss of urine involuntary and combined by urgency) and mixed UI (MUI) (combination of the two). UUI is the second most common type of UI in women, and it is estimated that 20-40% of women who visit outpatient clinic healthcare services have UUI. Regarding women with SUI, the surgical intervention by using a tension free vaginal tape is a successful method. Considering females with UUI, the pharmacological treatment is a long-lasting and effective alternative.

Pathophysiology of overactive bladder in women with POP Few evidence exist regarding the etiology of OAB in women with POP. POP itself is considered an important mechanism for the development of OAB. Several studies have suggested that patients with POP have a lower peak of maximum flow rate (Q max) during urination compared to patients without concomitant prolapse. In addition, the average flow rate (Q ave) in women with detrusor overactivity appears to be lower as well. It is possible that obstructive urination is involved in the creation of the detrusor overactivity in patients with POP . In studies with patients who underwent POP surgery, had improvement of OAB symptoms, and the urinary flow rates were mainly improved postoperatively.

The first theory that attempts to explain how prolapse induces the OAB symptoms is the possible damage of bladder nerve pathways that happens in women with obstructive voiding. In these patients, hypersensitivity and decreased secretion of acetylcholine (Ach), which is the major neurotransmitter of the urinary bladder, was found in comparison to asymptomatic patients. Ischemia and bladder wall hypoxia caused by bladder dilatation and contractions may play an important role in this damaged neural pathway in cases of prolapse and obstructive urination.

The second theory focuses on the bladder detrusor muscle. The urinary bladder is a hollow sac-like cavity connected with the ureters, where the urine is collected, and a funnel extension, the bladder neck connected to the urethra. The urinary bladder is lined with transitional epithelial tissue that is able to stretch significantly to accommodate large volumes of urine. The main part of the wall is formed by smooth muscle layers provide the urinary bladder with its ability to expand and contract. It is commonly referred to as the detrusor muscle. In cases where there is a reduction in the cell-site electrical activity propagation or in the cell membrane instability, the transmission of the cell-to-cell electrical activity signal is activated. As a result, the detrusor muscle becomes hypersensitive and the patient develops OAB symptoms.

According to the third theory, changes in the spinal reflexes are the cause of the OAB. In experimental animal studies, bladder obstruction has been shown to cause hypertrophy of the afferent neurons and is accompanied by increased expression of NGF in the bladder wall. Also, it was shown that obstruction is accompanied to a certain extent by a reduction in neuronal excitability leading to a more pronounced spinal reflex that could contribute to the development of OAB.

Other possible pathophysiological mechanisms of OAB in women suffering from POP is the dilatation of the bladder wall, which commonly appears in POP and which can induce receptor stimulation resulting in contractions of the detrusor muscle Finally, a large sized vaginal prolapse can drop down the bladder neck and the most common symptom is UI. This mechanism is known to cause detrusor overactivity (DO).

The role of biomarkers in the diagnosis and monitoring of overactive bladder A. The bladder wall thickness (BWT) There are numerous studies linking the increase in bladder wall thickness (BWT) with the symptoms of the OAB. It appears that BWT is affected by the increased muscle work that occurs due to DO. In several studies, ultrasound transvaginal scanning of the detrusor muscle over 5mm is significantly associated with OAB symptomatology. Finally, there is little evidence of altering the BWT in women with OAB after treatment with anticholinergics. To conclude, there are no studies to investigate BWT in women with POP and OAB symptoms.

B. Neurotrophic Growth Factor (NGF) Neurotrophins are responsible for the maintenance and the control of bladder nerve stimulation threshold and appear to be involved in the pathophysiology of the OAB symptoms. NGF is produced by urothelium and smooth muscles of the detrusor muscle and its urine levels seems to rise in OAB patients and to fall after a successful treatment. In studies where the objective was to investigate the role of NGF in the pathophysiology of lower urinary tract symptoms, it was found that urinary NGF levels were consistently low in asymptomatic women. In similar studies in patients with lower urinary tract symptoms, urinary NGF levels were found to be elevated. Finally, in studies in which the symptoms of OAB were successfully treated, urinary NGF levels were reduced. There are also no studies to investigate urinary NGF levels in women with prolapse and coexisting bladder symptomatology.

Are symptoms of OAB improved after treatment for POP? In literature, there are still no sufficient high quality studies to address this question. There is only one study with Stage I prolapse patients and a smaller group with Stage II prolapse, all of which had proven symptoms of OAB and urodynamically documented DO. After conservative pharmacological treatment with tolterodine, only 14.1% of Stage I patients and 39.2% of Stage II patients continued to experience OAB symptoms. This study showed an improvement in OAB in patients with vaginal prolapse (relative risk-RR) of 2.55, but improvement in women without prolapse was much higher (RR 7.09). The difference could be explained in some extent because of the fact that OAB is provoked by vaginal prolapse itself and continues to exist despite conservative treatment. In the other hand, there are more than 12 studies in the literature showing that symptoms of OAB are improved after surgical treatment for vaginal prolapse, including de novo overactive bladder postoperatively.

Detrusor overactivity (DO) The presence of vaginal prolapse appears to be a risk factor for the DO, since in urodynamic studies appear to co-exist at a rate of 10-50%. The majority of studies show improvement of DO activity after surgical repair of vaginal prolapse. Overall, it appears that there is a high probability of disappearance of DO after surgery, but these results do not seem to be verified in cases of concomitant OAB.

In summary, there is a large number of women suffering from POP and UI problems. There is the possibility to repair surgically both conditions in case of SUI with high rates of success. In case of UUI, the surgical repair of vaginal prolapse shows up to 50% improvement in UI postoperatively. However, it is not yet investigated whether there are some specific biomarkers that could help to assess and predict patients with POP and UUI who would be benefit by a surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult women that are able to communicate and understand comprehensively Greek Language and present vaginal prolapse problems.

Exclusion Criteria:

* Male patients as well children will be excluded.
* Women that have already operated once for pelvic organ prolapse.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women that visited outpatients Gynecology Department, 1st Department Obstetrics and Gynecology, Aristotle University of Thessaloniki, General Hospital Papageorgiou of Thessaloniki, complaining for vaginal prolapse and possible concomitant urinary problems.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2018-01-29 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Urinary NGF as a biomarker for OAB symptoms in women with POP | Two samples will be taken at the time of recruitment (Month 0) at three months post-operatively (Month 3).
  Determination of urinary NGF levels' change as a reliable prognostic factor for the treatment of OAB in women with POP before and after surgical repair
Urinary NGF as a biomarker for OAB symptoms in women with POP | Two samples will be taken at the time of recruitment (Month 0) and at the 1 years follow up appointment post-operatively (Month 12)
  Determination of urinary NGF levels' change as a reliable prognostic factor for the treatment of OAB in women with POP before and after surgical repair.

SECONDARY OUTCOMES:
BWT as a biomarker for OAB symptoms in women with POP | Ultrasound will take place before surgery repair (Month 0) at three months post-operatively (Month 3).
  Determination of BWT's change as a reliable prognostic factor for the treatment of OAB in women with POP.

CONTACTS AND LOCATIONS:
Overall Officials: Themistoklis Mikos, MD PhD, Study Director — Aristotle University Of Thessaloniki
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, Central Macedonia, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Boer TA, Salvatore S, Cardozo L, Chapple C, Kelleher C, van Kerrebroeck P, Kirby MG, Koelbl H, Espuna-Pons M, Milsom I, Tubaro A, Wagg A, Vierhout ME. Pelvic organ prolapse and overactive bladder. Neurourol Urodyn. 2010;29(1):30-9. doi: 10.1002/nau.20858. PMID 20025017
- [Background] de Boer TA, Kluivers KB, Withagen MI, Milani AL, Vierhout ME. Predictive factors for overactive bladder symptoms after pelvic organ prolapse surgery. Int Urogynecol J. 2010 Sep;21(9):1143-9. doi: 10.1007/s00192-010-1152-y. Epub 2010 Apr 24. PMID 20419366
- [Background] Rachaneni S, McCooty S, Middleton LJ, Parker VL, Daniels JP, Coomarasamy A, Verghese TS, Balogun M, Goranitis I, Barton P, Roberts TE, Deeks JJ, Latthe P; Bladder Ultrasound Study (BUS) Collaborative Group. Bladder ultrasonography for diagnosing detrusor overactivity: test accuracy study and economic evaluation. Health Technol Assess. 2016 Jan;20(7):1-150. doi: 10.3310/hta20070. PMID 26806032
- [Background] Seth JH, Sahai A, Khan MS, van der Aa F, de Ridder D, Panicker JN, Dasgupta P, Fowler CJ. Nerve growth factor (NGF): a potential urinary biomarker for overactive bladder syndrome (OAB)? BJU Int. 2013 Mar;111(3):372-80. doi: 10.1111/j.1464-410X.2012.11672.x. PMID 23444927
- [Background] Wu JM, Matthews CA, Conover MM, Pate V, Jonsson Funk M. Lifetime risk of stress urinary incontinence or pelvic organ prolapse surgery. Obstet Gynecol. 2014 Jun;123(6):1201-1206. doi: 10.1097/AOG.0000000000000286. PMID 24807341
- [Background] Forde JC, Davila JL, Marks BK, Epstein M, Tsui JF, Weiss JP, Blaivas JG. Urogynecological conditions associated with overactive bladder symptoms in women. Can Urol Assoc J. 2017 Mar-Apr;11(3-4):E83-E87. doi: 10.5489/cuaj.3962. Epub 2017 Mar 16. PMID 28360952
- [Background] Eapen RS, Radomski SB. Review of the epidemiology of overactive bladder. Res Rep Urol. 2016 Jun 6;8:71-6. doi: 10.2147/RRU.S102441. eCollection 2016. PMID 27350947
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Background] Bureau M, Carlson KV. Pelvic organ prolapse: A primer for urologists. Can Urol Assoc J. 2017 Jun;11(6Suppl2):S125-S130. doi: 10.5489/cuaj.4634. PMID 28616110
- [Background] Osman T. Stress incontinence surgery for patients presenting with mixed incontinence and a normal cystometrogram. BJU Int. 2003 Dec;92(9):964-8. doi: 10.1111/j.1464-410x.2003.04519.x. PMID 14632856
- [Background] Olivera CK, Meriwether K, El-Nashar S, Grimes CL, Chen CC, Orejuela F, Antosh D, Gleason J, Kim-Fine S, Wheeler T, McFadden B, Balk EM, Murphy M; Systematic Review Group for the Society of Gynecological Surgeons. Nonantimuscarinic treatment for overactive bladder: a systematic review. Am J Obstet Gynecol. 2016 Jul;215(1):34-57. doi: 10.1016/j.ajog.2016.01.156. Epub 2016 Feb 4. PMID 26851599
- [Background] Zargham M, Alizadeh F, Moayednia A, Haghdani S, Nouri-Mahdavi K. The role of pelvic organs prolapse in the etiology of urinary incontinence in women. Adv Biomed Res. 2013 Mar 6;2:22. doi: 10.4103/2277-9175.108010. eCollection 2013. PMID 23977650
- [Background] Long CY, Hsu SC, Sun DJ, Chen CC, Tsai EM, Su JH. Abnormal clinical and urodynamic findings in women with severe genitourinary prolapse. Kaohsiung J Med Sci. 2002 Dec;18(12):593-7. PMID 12670034
- [Background] Rosenzweig BA, Pushkin S, Blumenfeld D, Bhatia NN. Prevalence of abnormal urodynamic test results in continent women with severe genitourinary prolapse. Obstet Gynecol. 1992 Apr;79(4):539-42. PMID 1553172
- [Background] Coates KW, Harris RL, Cundiff GW, Bump RC. Uroflowmetry in women with urinary incontinence and pelvic organ prolapse. Br J Urol. 1997 Aug;80(2):217-21. doi: 10.1046/j.1464-410x.1997.00246.x. PMID 9284191
- [Background] Basu M, Duckett J. Effect of prolapse repair on voiding and the relationship to overactive bladder and detrusor overactivity. Int Urogynecol J Pelvic Floor Dysfunct. 2009 May;20(5):499-504. doi: 10.1007/s00192-009-0807-z. Epub 2009 Feb 12. PMID 19214362
- [Background] Salvatore S, Serati M, Ghezzi F, Uccella S, Cromi A, Bolis P. Efficacy of tolterodine in women with detrusor overactivity and anterior vaginal wall prolapse: is it the same? BJOG. 2007 Nov;114(11):1436-8. doi: 10.1111/j.1471-0528.2007.01399.x. Epub 2007 Sep 17. PMID 17877779
- [Background] Azadzoi KM, Pontari M, Vlachiotis J, Siroky MB. Canine bladder blood flow and oxygenation: changes induced by filling, contraction and outlet obstruction. J Urol. 1996 Apr;155(4):1459-65. doi: 10.1016/s0022-5347(01)66307-9. PMID 8632611
- [Background] Gosling JA, Gilpin SA, Dixon JS, Gilpin CJ. Decrease in the autonomic innervation of human detrusor muscle in outflow obstruction. J Urol. 1986 Aug;136(2):501-4. doi: 10.1016/s0022-5347(17)44930-5. PMID 3735523
- [Background] van Koeveringe GA, Mostwin JL, van Mastrigt R, van Koeveringe BJ. Effect of partial urethral obstruction on force development of the guinea pig bladder. Neurourol Urodyn. 1993;12(6):555-66; discussion 566-71. doi: 10.1002/nau.1930120607. PMID 8312940
- [Background] Steers WD, Kolbeck S, Creedon D, Tuttle JB. Nerve growth factor in the urinary bladder of the adult regulates neuronal form and function. J Clin Invest. 1991 Nov;88(5):1709-15. doi: 10.1172/JCI115488. PMID 1939656
- [Background] Steers WD, Ciambotti J, Etzel B, Erdman S, de Groat WC. Alterations in afferent pathways from the urinary bladder of the rat in response to partial urethral obstruction. J Comp Neurol. 1991 Aug 15;310(3):401-10. doi: 10.1002/cne.903100309. PMID 1723990
- [Background] Ferguson DR, Kennedy I, Burton TJ. ATP is released from rabbit urinary bladder epithelial cells by hydrostatic pressure changes--a possible sensory mechanism? J Physiol. 1997 Dec 1;505 ( Pt 2)(Pt 2):503-11. doi: 10.1111/j.1469-7793.1997.503bb.x. PMID 9423189
- [Background] Yoshida M, Masunaga K, Satoji Y, Maeda Y, Nagata T, Inadome A. Basic and clinical aspects of non-neuronal acetylcholine: expression of non-neuronal acetylcholine in urothelium and its clinical significance. J Pharmacol Sci. 2008 Feb;106(2):193-8. doi: 10.1254/jphs.fm0070115. Epub 2008 Feb 16. PMID 18285653
- [Background] Jung SY, Fraser MO, Ozawa H, Yokoyama O, Yoshiyama M, De Groat WC, Chancellor MB. Urethral afferent nerve activity affects the micturition reflex; implication for the relationship between stress incontinence and detrusor instability. J Urol. 1999 Jul;162(1):204-12. doi: 10.1097/00005392-199907000-00069. PMID 10379788
- [Background] Serati M, Salvatore S, Cattoni E, Soligo M, Cromi A, Ghezzi F. Ultrasound measurement of bladder wall thickness in different forms of detrusor overactivity. Int Urogynecol J. 2010 Nov;21(11):1405-11. doi: 10.1007/s00192-010-1194-1. Epub 2010 Jun 10. PMID 20535449
- [Background] Panayi DC, Tekkis P, Fernando R, Khullar V. Is the beneficial effect of antimuscarinics related to motor or sensory changes in the bladder? Int Urogynecol J. 2010 Jul;21(7):841-5. doi: 10.1007/s00192-010-1123-3. Epub 2010 Mar 27. PMID 20349178
- [Background] Cruz F, Heesakkers J, Khullar V, Tubaro A. Bladder Wall Thickness in Overactive Bladder: Does It Have a Role? Eur Urol Suppl. 2009; 8(9):769-71
- [Background] Antunes-Lopes T, Cruz CD, Cruz F, Sievert KD. Biomarkers in lower urinary tract symptoms/overactive bladder: a critical overview. Curr Opin Urol. 2014 Jul;24(4):352-7. doi: 10.1097/MOU.0000000000000064. PMID 24841379
- [Background] Schaefer W. Comment on Kuo: Measurement of detrusor wall thickness in women with overactive bladder by transvaginal and transabdominal sonography. Int Urogynecol J. 2010 Jan;21(1):129-30; author reply 131-2. doi: 10.1007/s00192-009-0999-2. Epub 2009 Sep 29. No abstract available. PMID 19787280
- [Background] Blatt AH, Titus J, Chan L. Ultrasound measurement of bladder wall thickness in the assessment of voiding dysfunction. J Urol. 2008 Jun;179(6):2275-8; discussion 2278-9. doi: 10.1016/j.juro.2008.01.118. Epub 2008 Apr 18. PMID 18423703
- [Background] Robinson D, Oelke M, Khullar V, Wijkstra H, Tretter R, Stow B, Compion G, Tubaro A. Bladder wall thickness in women with symptoms of overactive bladder and detrusor overactivity: Results from the randomised, placebo-controlled shrink study. Neurourol Urodyn. 2016 Sep;35(7):819-25. doi: 10.1002/nau.22808. Epub 2015 Jul 21. PMID 26199198
- [Background] Cruz CD. Neurotrophins in bladder function: what do we know and where do we go from here? Neurourol Urodyn. 2014 Jan;33(1):39-45. doi: 10.1002/nau.22438. Epub 2013 Jun 17. PMID 23775873
- [Background] Liu HT, Kuo HC. Urinary nerve growth factor level could be a potential biomarker for diagnosis of overactive bladder. J Urol. 2008 Jun;179(6):2270-4. doi: 10.1016/j.juro.2008.01.146. Epub 2008 Apr 18. PMID 18423678
- [Background] Liu HT, Chancellor MB, Kuo HC. Urinary nerve growth factor levels are elevated in patients with detrusor overactivity and decreased in responders to detrusor botulinum toxin-A injection. Eur Urol. 2009 Oct;56(4):700-6. doi: 10.1016/j.eururo.2008.04.037. Epub 2008 Apr 30. PMID 18472208
- [Background] Kuo HC, Liu HT, Chancellor MB. Can urinary nerve growth factor be a biomarker for overactive bladder? Rev Urol. 2010 Spring;12(2-3):e69-77. PMID 20811555
- [Background] Liu HT, Chancellor MB, Kuo HC. Decrease of urinary nerve growth factor levels after antimuscarinic therapy in patients with overactive bladder. BJU Int. 2009 Jun;103(12):1668-72. doi: 10.1111/j.1464-410X.2009.08380.x. Epub 2009 Feb 11. PMID 19220267
- [Background] Bray R, Cartwright R, Cardozo L, Hill S, Guan Z, Khullar V. Tolterodine ER reduced increased bladder wall thickness in women with overactive bladder. A randomized, placebo-controlled, double-blind, parallel group study. Neurourol Urodyn. 2018 Jan;37(1):237-243. doi: 10.1002/nau.23281. Epub 2017 Apr 13. PMID 28407338
- [Background] Digesu GA, Salvatore S, Chaliha C, Athanasiou S, Milani R, Khullar V. Do overactive bladder symptoms improve after repair of anterior vaginal wall prolapse? Int Urogynecol J Pelvic Floor Dysfunct. 2007 Dec;18(12):1439-43. doi: 10.1007/s00192-007-0375-z. Epub 2007 Apr 11. PMID 17429557
- [Background] Brubaker L, Cundiff GW, Fine P, Nygaard I, Richter HE, Visco AG, Zyczynski H, Brown MB, Weber AM; Pelvic Floor Disorders Network. Abdominal sacrocolpopexy with Burch colposuspension to reduce urinary stress incontinence. N Engl J Med. 2006 Apr 13;354(15):1557-66. doi: 10.1056/NEJMoa054208. PMID 16611949
- [Background] Lekskulchai O, Dietz HP. Detrusor wall thickness as a test for detrusor overactivity in women. Ultrasound Obstet Gynecol. 2008 Sep;32(4):535-9. doi: 10.1002/uog.5370. PMID 18634113
- [Background] Liang CC, Tseng LH, Chang YL, Chang SD. Predictors of persistence of preoperative urgency incontinence in women following pelvic organ prolapse repair. Taiwan J Obstet Gynecol. 2015 Dec;54(6):682-5. doi: 10.1016/j.tjog.2014.08.012. PMID 26700985
- [Background] Weber AM, Walters MD, Piedmonte MR, Ballard LA. Anterior colporrhaphy: a randomized trial of three surgical techniques. Am J Obstet Gynecol. 2001 Dec;185(6):1299-304; discussion 1304-6. doi: 10.1067/mob.2001.119081. PMID 11744900